CLINICAL TRIAL: NCT07294833
Title: Investigation of Respiratory Functions, Respiratory Muscle Strength, Balance and Sleep Quality in Patients With Bruxism
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: Gazi2710
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Bruxism; Respiratory Function; Sleep Quality; Balance
Keywords: bruxism; respiratory functions; respiratory muscle strength; balance; sleep quality
MeSH Terms: conditions — Bruxism; Respiratory Aspiration; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with bruxism: Information about the diagnostic required for the study, type of bruxism, duration of symptoms, duration of diagnosis were recorded from the patient's files. All assessments were performed once, in a temperature-controlled, quiet laboratory setting, by experienced physiotherapists. The evaluated parameters included pulmonary function, respiratory muscle strength, balance performance, and sleep quality.
- Health Controls: All assessments were performed once, in a temperature-controlled, quiet laboratory setting, by experienced physiotherapists. The evaluated parameters included pulmonary function, respiratory muscle strength, balance performance, and sleep quality.

SUMMARY:
It has been reported that patients with bruxism frequently present with upper respiratory tract symptoms such as rhinitis, sinusitis, and mouth breathing. Upper respiratory tract infections have been shown to reduce lung volumes, and individuals with bruxism commonly exhibit forward head posture, which is known to negatively affect postural balance. However, no studies have investigated respiratory function or respiratory muscle strength in patients with bruxism, and the number of studies evaluating balance in this population is limited. The aim of the present study is to assess respiratory function, respiratory muscle strength, balance, and sleep quality in individuals with bruxism and to compare these outcomes with those of healthy controls.

DETAILED DESCRIPTION:
Bruxism is defined as an involuntary, irregular, or rhythmic parafunctional oral activity characterized by clenching or grinding of the teeth, without serving any functional chewing purpose. Various central, pathophysiological, psychosocial, morphological, environmental, and biological factors have been proposed in the etiology of sleep bruxism. Three subtypes of bruxism are described: awake (diurnal) bruxism, which occurs during wakefulness; sleep (nocturnal) bruxism, which occurs during sleep; and combined bruxism, in which features of both are present. Common symptoms include temporomandibular joint pain, discomfort in the masticatory and cervical muscles, headaches-particularly in the temporal region-poor sleep quality, fatigue, and recurrent migraine attacks. Increasing evidence suggests that respiration plays a notable role in the pathophysiology of sleep bruxism. Researchers have reported specific alterations in breathing patterns among affected individuals, proposing that sleep is often associated with a mandibular open or retruded position, which may lead to reduced airway patency due to relaxation of the tongue muscles. It has also been suggested that sleep bruxism may be associated with reduced airway flow or increased upper airway resistance, particularly in individuals who tend to sleep in the supine position.

Clinicians are encouraged to consider the coexistence of sleep-related breathing disturbances-such as snoring, upper airway resistance, or apnea-hypopnea-in patients presenting with sleep bruxism. Snoring, the most common initial respiratory disturbance during sleep, is defined as an oropharyngeal sound resulting from turbulent airflow that causes vibration of soft tissues. In addition, patients with bruxism frequently experience symptoms associated with upper respiratory tract involvement, including rhinitis, sinusitis, and mouth breathing. Upper respiratory tract infections have been shown to reduce lung volumes, and mouth breathing is thought to influence cerebral oxygenation and provoke involuntary contractions of the facial musculature, potentially triggering sleep bruxism. Despite these associations, no studies to date have investigated pulmonary function or respiratory muscle strength in individuals with bruxism.

Bruxism is also associated with dental damage, temporomandibular joint dysfunction, headaches, and postural alterations. These findings indicate that bruxism affects not only the masticatory muscles but also the craniofacial complex and the musculature of the neck and shoulders. Previous studies have demonstrated that individuals with bruxism, particularly children, exhibit a more pronounced forward head posture compared with non-bruxism controls. A forward shift of the head increases the mechanical load on the cervical region and can alter the body's center of gravity, potentially contributing to muscular imbalance and impairments in postural stability. Thus, head posture should be considered in the clinical evaluation of bruxism. Although balance has been examined in individuals with temporomandibular joint dysfunction, studies focusing specifically on balance in patients with bruxism are lacking, and research including bruxism populations within broader temporomandibular dysfunction cohorts remains limited.

Sleep is a vital physiological process during which sensory perception and neuromuscular function are restored and hormonal rhythms are regulated. It consists of multiple stages that differ physiologically and interact with circadian mechanisms to regulate the sleep-wake cycle. When sleep is disrupted-by sleep bruxism, chronic insomnia, narcolepsy, sleep apnea, or other disorders-functional alterations in sleep architecture may occur, negatively affecting quality of life and contributing to public health concerns. Despite the known associations between bruxism, respiratory disturbances, postural alterations, and sleep disruption, no studies have investigated respiratory muscle strength or pulmonary function specifically in individuals with bruxism, and only a few studies have evaluated balance in this population.

The aim of the present study is to assess respiratory muscle strength, respiratory function, balance, and sleep quality in individuals with bruxism using valid, reliable, and objective measurement methods, and to compare these findings with those of healthy controls. This work seeks to address important gaps in the literature and contribute novel insights into the multisystem effects of bruxism.

ELIGIBILITY:
Inclusion Criteria (bruxism group):

* Aged 18-65 years.
* Diagnosed with sleep or awake bruxism by a dentomaxillofacial radiologist.
* Diagnosis was based on subjective reports and clinical assessment according to the Standardised Tool for the Assessment of Bruxism (STAB) framework.
* Classified as probable bruxism, defined as the presence of:
* Self-reported behaviors (e.g., grinding, clenching, bracing), and
* Clinical signs (e.g., tooth wear, linea alba, masseter hypertrophy).

Inclusion Criteria (healthy controls):

* Aged 18-65 years.
* Recruited through public campus advertisements.
* Matched for age and sex with the bruxism group.
* No history or symptoms of bruxism, confirmed by self-report and clinical examination.

Exclusion Criteria (applied to all participants):

* History of smoking.
* Respiratory conditions affecting pulmonary function (e.g., obstructive sleep apnea, chronic obstructive pulmonary disease, asthma).
* Difficulty understanding or following instructions.
* Presence of any dental or temporomandibular disorder other than bruxism.
* History of masseter botulinum toxin injection or facial/cervical trauma.
* Current use of sedatives, muscle relaxants, or centrally acting medications.
* Active orthodontic treatment.
* History of COVID-19 infection within the last six months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Seventeen individuals with bruxism and 17 healthy controls were compared.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | First day
  Pulmonary function was assessed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, forced expiratory volume in the first second (FEV1) was assessed.
Pulmonary function (Forced vital capacity (FVC)) | First Day
  Pulmonary function was assesed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, forced vital capacity (FVC) was assessed
Pulmonary function (FEV1 / FVC) | First Day
  Pulmonary function was assessed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, FEV1 / FVC was assessed.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | First Day
  Pulmonary function was assessed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) was assessed
Pulmonary function (Peak flow rate (PEF)) | First Day
  Pulmonary function was assessed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, peak flow rate (PEF) was assessed.
Respiratory Muscle Strength | First day
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength were measured using a portable mouth pressure measuring device according to American Thoracic Society and European Respiratory Society criteria

SECONDARY OUTCOMES:
Posture assessment | First Day
  Posture assessment form of Corbin et al. was used for posture assessment. The form provides scoring according to the severity of postural disorders observed from lateral and posterior (0=absent, 1=mild, 2=moderate, 3=severe).
Balance | First Day
  Balance was assessed with the Y balance test. Participants were asked to stand on the central junction point of 3 tape measures; each fixed to the ground at 120-degree angles.
Sleep quality | First Day
  Sleep quality was assessed with the Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 24 questions, and these questions are also evaluated as 7 components. Each question is scored according to the values of the numbers from 0 to 3, and the total score is obtained by adding the scores of the 7 components.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Yoleri, MSc, Study Chair — Gazi University; Meral Boşnak Güçlü, Prof, Study Director — Gazi University; Musa Güneş, PhD, Principal Investigator — Karabük University; Nebiha Gözde İspir, MD, Principal Investigator — Gazi University; Okan Karaoğlu, Pt, Principal Investigator — Gazi University; Dilek Kaya, Pt, Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Cardiopulmonary Physiotherapy and Rehabilitation, Ankara, Çankaya 06490, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Castroflorio T, Bargellini A, Rossini G, Cugliari G, Deregibus A. Sleep bruxism in adolescents: a systematic literature review of related risk factors. Eur J Orthod. 2017 Feb;39(1):61-68. doi: 10.1093/ejo/cjw012. Epub 2016 Feb 15. PMID 26884421
- [Result] Manfredini D, Bucci MB, Sabattini VB, Lobbezoo F. Bruxism: overview of current knowledge and suggestions for dental implants planning. Cranio. 2011 Oct;29(4):304-12. doi: 10.1179/crn.2011.045. PMID 22128671
- [Result] Cuccia A, Caradonna C. The relationship between the stomatognathic system and body posture. Clinics (Sao Paulo). 2009;64(1):61-6. doi: 10.1590/s1807-59322009000100011. PMID 19142553
- [Result] Fabozzi A, Steffanina A, Nicolai A, Olmati F, Bonini M, Palange P. The Impact of Lung Function on Sleep Monitoring in Obstructive Sleep Apnea Associated with Obstructive Lung Diseases: Insights from a Clinical Study. J Clin Med. 2024 Oct 17;13(20):6189. doi: 10.3390/jcm13206189. PMID 39458139
- [Result] Shaffer SW, Teyhen DS, Lorenson CL, Warren RL, Koreerat CM, Straseske CA, Childs JD. Y-balance test: a reliability study involving multiple raters. Mil Med. 2013 Nov;178(11):1264-70. doi: 10.7205/MILMED-D-13-00222. PMID 24183777
- [Result] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Result] Johnson JD, Theurer WM. A stepwise approach to the interpretation of pulmonary function tests. Am Fam Physician. 2014 Mar 1;89(5):359-66. PMID 24695507